CLINICAL TRIAL: NCT00614926
Title: Modafinil for Treatment of Fatigue in ALS Patients: Pilot Study
Brief Title: Modafinil for Treatment of Fatigue in ALS Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5178
Record Dates: First submitted 2007-12-28; First posted 2008-02-13 (Estimated); Results first posted 2011-07-25 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Fatigue
Keywords: Fatigue; low energy; ALS; treatment
MeSH Terms: conditions — Fatigue | interventions — Modafinil; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Modafinil (Experimental): Eligible patients will be treated at baseline through Week 4. Those who choose to continue will have additional in-person visits at Weeks 8 and 12 visits (and Week 16 for those starting modafinil at Week 4).
  Interventions: Drug: Modafinil
- Placebo (Placebo Comparator): Sugar pill equivalent to the active comparator. Dosing schedule will be the same as the dosing schedule for Modafinil.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Modafinil — Dose schedule: 50 mg/day for 1 week, increasing to 100 mg/day at Week 2. Thereafter, dose may be increased to 300 mg/day as clinically indicated, in the absence of dose-limiting side effects. Dose is daily, in A.M., for 4 weeks.
  Other Names: Provigil
  Arms: Modafinil
Drug: Placebo — Placebo capsules are administered on the same schedule as active drug: 50 mg/day for 1 week, increasing to 100 mg/day at Week 2. Thereafter, dose may be increased to 300 mg/day in the absence of clinical improvement and dose limiting side effects. Dose is daily, in A.M.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
The purpose of this pilot study is to evaluate whether modafinil is helpful in alleviating fatigue, low energy, drowsiness and difficulty concentrating among patients with amyotrophic lateral sclerosis (ALS), and to evaluate incidence and frequency of adverse events, if any.

DETAILED DESCRIPTION:
ALS is an untreatable, progressive, fatal neurodegenerative disease whose etiology is unknown and whose course is relatively rapid (median survival 3 years after diagnosis). Palliative care, including symptom management, can contribute greatly to improved quality of life. In this context, alleviation of fatigue can help maintain function, extend the duration of time when employment is feasible for those still working, and can enable patients to more fully participate in and enjoy social and recreational activities. Given the prevalence of fatigue in this population, identification of effective treatment is a meaningful goal.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ALS
* Ages 18-80
* Clinically significant fatigue (4.5+ on Fatigue Severity Scale with duration 3+ months plus impairment in 1+ categories of role function)
* Speaks English
* Able and willing to give informed consent
* Can communicate verbally or with assistive device
* Can swallow capsules
* Forced vital capacity 50+%

Exclusion Criteria:

* Untreated hypothyroidism (TSH > 4.25 UIU/ML)
* Untreated and uncontrolled hypertension
* Clinically significant anemia (HCT < 33%)
* Untreated or under-treated major depressive disorder
* Current clinically significant suicidal ideation
* Started antidepressant medication for treatment of depression during past 6 weeks
* Currently taking psychostimulant medication
* History or current psychosis or bipolar disorder
* Fecund women not currently using barrier methods of contraception

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith G Rabkin, PhD, Principal Investigator — professor
Locations (1):
- New York State Psychiatric Institute-Columbia University, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: dates of recruitment were June 2006 through October 2007 at at the MDA-ALS Neurology Clinic at Columbia University.
Pre-assignment Details: Medical exclusion criteria were low thyroid levels which led to 3 patients excluded.
Period: Overall Study
Arm/Group | Modafinil | Placebo
Started | 25 | 7
Completed | 21 | 7
Not Completed | 4 | 0
Not completed — Burden of travel | 1 | 0
Not completed — Adverse Event | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Modafinil | Placebo | Total
Number analyzed (Participants) | 25 | 7 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 6 | 29
  >=65 years | 2 | 1 | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 59 (13) | 56 (5) | 58 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 3 | 14
  Male | 14 | 4 | 18
Region of Enrollment [Number; unit: participants]
  United States | 25 | 7 | 32
Fatigue Severity Scale score >40 [Number; unit: participants] — Minimum score = 9, maximum = 63. Nine items, no subscales. Higher scores signify greater fatigue. Total summed scores over 40 (equal to mean item score of 4.5+) are considered to signify "clinically significant fatigue" and was a requirement for study eligibility.
  participants | 25 | 7 | 32

OUTCOME MEASURES:

1. Primary Outcome: Participants Considered "Responders" (Scored 1 or 2) on Clinical Global Impressions Scale
Description: The CGI is a standardized assessment tool widely used in clinical psychopharmacology trials as an outcome measure. Scores range from 1= very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5-7 = worse. We use it as a dichotomous measure with scores of 1 or 2 signifying "responder" and all the rest as "non-responder" using all available data including clinician judgement, and ratings scales.
Time Frame: 4 weeks
Population: Analysis was Intention to Treat (ITT) including Last-Observation-Carried-Forward (LOCF) as indicated. Proof of concept study so N was based on accrual feasibility.
Measure: Number; unit: participants considered "responders"
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 25 | 7
participants considered "responders" | 19 | 1

2. Secondary Outcome: Number of "Impaired" Scores on Neuropsychological (Brief) Test Battery
Description: This was an initial plan but the large majority of patients were too impaired (either anarthric or unable to use hands) to complete the tests we had selected so this outcome measure turned out to be unfeasible. Therefore, 0 participants were analyzed.
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Modafinil | Placebo
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/7
Other Adverse Events (participants affected / at risk) | 0/25 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes